CLINICAL TRIAL: NCT01862146
Title: Response-to-injury in Patients Undergoing Transradial Coronary Angiography: Arterial Remodeling in Smokers
Brief Title: Arterial Remodeling in Smokers
Acronym: TCA
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: TCA INJURY
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: FMD; IMT; Smoking
Keywords: TCA; FMD; IMT; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Current Smoker underwent TCA: subjects who smokes daily
  Interventions: Procedure: smoke expose
- Former Smokers underwent TCA: subjects who do not smoke since 7 years

INTERVENTIONS:
Procedure: smoke expose
  Groups: Current Smoker underwent TCA

SUMMARY:
Cigarette smoking is the most important modifiable cardiovascular risk factor leading to endothelial dysfunction and was suggested to impair arterial regeneration.The aim of the study was to investigate the effect of smoking on vascular response to transradial coronary angiography (TCA).

ELIGIBILITY:
Inclusion Criteria:

* all subjects underwent a TCA

Exclusion Criteria:

* acute inflammation cardiac arrhythmia renal failure heart failure (NYHA II-IV) CRP > 1 mg/dl malignant disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all subjects who underwent an TCA (trans radial catheterisation)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
IMT hyperplasia | change in radials IMT after 6-14 month after a TCA
  IMT is measured by high resolution ultrasound in the radial arteries.

SECONDARY OUTCOMES:
Endothelial function | change in flow mediated dilatation after 10-14 months
  Flow mediated dilatation (FMD)

OTHER OUTCOMES:
cell migration | baseline
  measured by boyden chamber from blood plasma
Regeneration | baseline
  measured by scratch assay

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine Duesseldorf,, Düsseldorf, North Rhine-Westphalia, Germany